CLINICAL TRIAL: NCT03292133
Title: A Phase 2 Study of EGF816 and Gefitinib in TKI-naïve EGFR-mutant Non-Small Cell Lung Cancer
Brief Title: A Study of EGF816 and Gefitinib in TKI-naïve EGFR-mutant Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Zofia Piotrowska, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-291
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — nazartinib; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EGF816 + Gefitinib (Experimental): * All patients will receive gefitinib orally once daily
  * EGF816 will be administered orally once daily
  * Participant will be requested to maintain a medication diary of each dose of medication
  Interventions: Drug: EGF816; Drug: Gefitinib

INTERVENTIONS:
Drug: EGF816 — EGF816 is an inhibitor which target a specific mutation in cancer and may stop tumors growing and multiplying
Drug: Gefitinib — Gefitinib is an inhibitor which target a specific mutation in cancer and may stop tumors growing and multiplying
  Other Names: Iressa

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for EGFR mutation-positive lung cancer.

The drugs involved in this study are:

* EGF816
* Gefitinib

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease or patient population. "Investigational" means that the drug or drugs are being studied and have not been approved together for patients.

The FDA (the U.S. Food and Drug Administration) has approved gefitinib as a treatment option for EGFR mutation-positive lung cancer.

The FDA has not approved EGF816 as a treatment for any disease at this time.

In this research study, the investigators are studying the safety and efficacy of the combination of the study drugs EGF816 and gefitinib.

Both EGF816 and gefitinib are inhibitors which target a specific mutation in cancer and may stop tumors growing and multiplying.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a pathologically-confirmed diagnosis of non-small cell lung cancer (NSCLC).
* Participants must have advanced disease - either stage IV disease, stage IIIB disease not amenable to definitive multi-modality therapy, or recurrent disease after a prior diagnosis of stage I-III disease. All staging is via the American Joint Committee on Cancer (AJCC)/IASLC 7th edition proposed staging criteria
* An EGFR sensitizing mutation must be detected in tumor tissue. Specifically, patients harboring the most common mutations, deletions in exon 19 or the L858R mutation in exon 21 are eligible. Other EGFR sensitizing mutations may be eligible after discussion with the principal investigator. Patients may be enrolled in the study based on an activating EGFR mutation detected by a CLIA-certified tissue or plasma-based assay, but will be required to undergo a mandatory tumor biopsy during study screening.
* Participants must have measurable disease, per RECIST 1.1. See Section 11 for the evaluation of measurable disease.
* Patients in the six patient safety run-in cohort may have had a prior EGFR TKI in the metastatic setting (to allow for patients who started initial therapy at an outside hospital), but treatment duration must have been less than three months. After the initial six-patient safety run-in, no prior EGFR TKI therapy in the metastatic setting is allowed. An EGFR TKI given in the adjuvant setting (i.e. with no measurable disease at the time of administration) is allowable provided the subject has been off of EGFR TKI therapy for at least six months at the time of enrollment.
* Patients may have had no more than one prior line of chemotherapy or immunotherapy in the metastatic setting. At least 14 days must have elapsed from the last chemo/immunotherapy administration until the start of protocol treatment, and patients must have recovered from the side effects of any of these agents.
* Patients must be screened for HBV. Patients who are either HBsAg positive or HBV-DNA positive must be willing and able to take antiviral therapy 1-2 weeks prior to 1st dose of study treatment and continue on antiviral therapy for at least 4 weeks after the last dose of EGF816. Additional management of the patients would be provided by a physician with expertise in management of HBV, if needed. Patients must have negative hepatitis C antibody (HCV-Ab) or positive HCV-Ab but undetectable level of HCV-RNA. Note: patients with detectable HCV-RNA are not eligible for the study.
* Patients must receive insurance approval for or be willing to pay for commercial gefitinib.
* Age >/= 18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Life expectancy of greater than 12 weeks.
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes ≥3,000/mcL
  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin >1.5 x upper limit of normal (ULN)

    *For patients with Gilbert's syndrome total bilirubin >3.0 x ULN
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal; for patients with known hepatic metastases AST and/or ALT > 5x ULN
  * Creatinine ≤1.5 × institutional upper limit of normal
* The effects of EGF816 and gefitinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use highly effective contraception during the study and for 3 months after stopping the study treatment. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptom thermal, postovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male Partner: male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
  * Combination of any two of the following (a+b or a+c, or b+c):
  * A. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
  * B. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
  * C. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
  * D. In case of use of oral contraception women should have been stable on the same pill for a minimum of 30 days before taking study treatment.
  * Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential.
  * Sexually active males must agree to use a condom during intercourse while taking drug and for 3 months after stopping treatment; men should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
* Ability to understand and the willingness to sign a written informed consent document. Written informed consent must be obtained prior to any screening procedures.

Exclusion Criteria:

* Participants with clinically active or symptomatic interstitial lung disease or interstitial pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention) and patients with history of clinically significant interstitial lung disease or radiation pneumonitis.
* Patients with clinically symptomatic brain metastases or leptomeningeal disease. Patients may be on a stable dose of corticosteroids to control brain metastases if they have been on a stable dose for two weeks prior to study treatment and are clinically asymptomatic.
* Patients who have had radiation to the lung fields within four weeks of starting treatment. For patients receiving palliative radiation to thoracic vertebrae, ribs or other sites where the radiation field includes the lungs, radiation must be completed at least two weeks before starting treatment. For all palliative radiation to all other sites, at least 7 days must have elapsed prior to starting to treatment. At least six months must have elapsed from radiation given with curative intent.
* Patients who have had major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 2 weeks prior to starting study drug or who have not recovered from side effects of such procedure. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and patients can be enrolled in the study ≥1 week after the procedure.
* Patients unable or unwilling to undergo a biopsy for research during the screening period, 2-3 weeks into the course of therapy and at the time of progression.
* Patients with a second, clinically active, cancer. Patients with second cancers which have been treated with curative intent and/or are currently inactive are allowed.
* Patients who have undergone a bone marrow or solid organ transplant.
* Known history of human immunodeficiency virus (HIV) seropositivity (HIV testing is not mandatory).
* Participants who are receiving any other investigational agents. Patients previously treated with investigational agents must complete a washout period of at least one week or five half-lives, whichever is longer, before starting treatment.
* Patients receiving concomitant immunosuppressive agents or chronic corticosteroid use, except those on steroid to control brain metastases, those on topical or inhaled steroids, or steroids given via local injection.
* Patients with clinically significant, uncontrolled cardiovascular disease, such as:

  * Unstable angina within 6 months prior to screening
  * Myocardial infarction within 6 months prior to screening
  * Patients with a history of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Peripheral vascular disease
  * Patients with uncontrolled hypertension defined as a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening
  * Ventricular arrhythmias
  * Supraventricular and nodal arrhythmias not controlled with medication
  * Other cardiac arrhythmia not controlled with medication
  * Patients with corrected QT (QTc) ≥450 ms (male patients) or ≥460 ms (female patients) using Fridericia correction (QTcF) on the screening ECG (using triplicate ECGs)
  * Patients with history of congenital long QT syndrome or history of torsade de pointes
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to EGF816 or gefitinib.
* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Unable or unwilling to swallow tablets or capsules.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because the effects of EGF816 and gefitinib on a developing fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with EGF816 or gefitinib, breastfeeding should be discontinued if the mother is treated with EGF816 and gefitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zofia Piotrowska, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EGF816 + Gefitinib: * All patients will receive gefitinib orally once daily
  * EGF816 will be administered orally once daily
  * Participant will be requested to maintain a medication diary of each dose of medication
  EGF816: EGF816 is an inhibitor which target a specific mutation in cancer and may stop tumors growing and multiplying
  Gefitinib: Gefitinib is an inhibitor which target a specific mutation in cancer and may stop tumors growing and multiplying
Period: Overall Study
Arm/Group | EGF816 + Gefitinib
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EGF816 + Gefitinib
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 58 [47 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: 9 Months Progression Free Rate
Description: The percentage of participants that are free from objective disease progression or death at 9 months after the start treatment. Progression is evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | EGF816 + Gefitinib
Number analyzed (Participants) | 11
Participants | 7

2. Secondary Outcome: Overall Response Rate (ORR)
Description: The number of participants that achieve either a complete response (CR) or a partial response (PR). Response is evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  All CRs and PRs must be confirmed by a second assessment not earlier than 4 weeks after the criteria for response are first met.
Time Frame: 4 years and 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | EGF816 + Gefitinib
Number analyzed (Participants) | 11
Participants | 8

3. Secondary Outcome: Median Overall Survival
Description: Overall survival is defined as time from the start of treatment until death or loss to follow up. Overall survival will be analyzed using the Kaplan-Meier method.
Time Frame: 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EGF816 + Gefitinib
Number analyzed (Participants) | 11
months | 35.7 [6.18 to NA] — Upper confidence interval not reached because too few survival events occurred.

4. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the time from start of treatment to the time of objective disease progression, death, or loss to follow up. Progression is evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 4.2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EGF816 + Gefitinib
Number analyzed (Participants) | 11
months | 20.86 [5.42 to 39.57]

5. Secondary Outcome: Summary of Treatment-related Adverse Events
Description: Treatment-related adverse events, defined as those at least possibly related to study treatment, are summarized below as a measure of patient safety and treatment tolerability. Subjects were evaluated for adverse events by the Common Terminology Criteria for Adverse Events (CTCAE) v4. For each treatment-related event, subjects are counted below by the highest grade they experienced on study per CTCAE v 4.0 to demonstrate the range and severity of treatment-related toxicities documented on study. Grade refers to the severity of the toxicity, with Grade 1 corresponding to mild toxicity, Grade 2 to moderate toxicity, and Grade 3 to severe toxicity. Patients who did not experience a given event at any grade are counted in the final category for each row.
Time Frame: Start of treatment through 30 days after the end of treatment (max 4 years and 5 months)
Measure: Count of Participants; unit: Participants
Arm/Group | EGF816 + Gefitinib
Number analyzed (Participants) | 11
Participants
  Anemia: Grade 1 (CTCAE v4) | 1
  Anemia: Grade 2 (CTCAE v4) | 0
  Anemia: Grade 3 (CTCAE v4) | 0
  Anemia: Subject did not experience this treatment-related toxicity | 10
  Cardiac disorders - other, specify: Grade 1 (CTCAE v4) | 0
  Cardiac disorders - other, specify: Grade 2 (CTCAE v4) | 1
  Cardiac disorders - other, specify: Grade 3 (CTCAE v4) | 0
  Cardiac disorders - other, specify: Subject did not experience this treatment-related toxicity | 10
  Dry eye: Grade 1 (CTCAE v4) | 1
  Dry eye: Grade 2 (CTCAE v4) | 0
  Dry eye: Grade 3 (CTCAE v4) | 0
  Dry eye: Subject did not experience this treatment-related toxicity | 10
  Eye Pain: Grade 1 (CTCAE v4) | 1
  Eye Pain: Grade 2 (CTCAE v4) | 0
  Eye Pain: Grade 3 (CTCAE v4) | 0
  Eye Pain: Subject did not experience this treatment-related toxicity | 10
  Abdominal Pain: Grade 1 (CTCAE v4) | 1
  Abdominal Pain: Grade 2 (CTCAE v4) | 0
  Abdominal Pain: Grade 3 (CTCAE v4) | 0
  Abdominal Pain: Subject did not experience this treatment-related toxicity | 10
  Bloating: Grade 1 (CTCAE v4) | 1
  Bloating: Grade 2 (CTCAE v4) | 0
  Bloating: Grade 3 (CTCAE v4) | 0
  Bloating: Subject did not experience this treatment-related toxicity | 10
  Diarrhea: Grade 1 (CTCAE v4) | 6
  Diarrhea: Grade 2 (CTCAE v4) | 3
  Diarrhea: Grade 3 (CTCAE v4) | 2
  Diarrhea: Subject did not experience this treatment-related toxicity | 0
  Dry mouth: Grade 1 (CTCAE v4) | 3
  Dry mouth: Grade 2 (CTCAE v4) | 0
  Dry mouth: Grade 3 (CTCAE v4) | 0
  Dry mouth: Subject did not experience this treatment-related toxicity | 8
  Dyspepsia: Grade 1 (CTCAE v4) | 1
  Dyspepsia: Grade 2 (CTCAE v4) | 0
  Dyspepsia: Grade 3 (CTCAE v4) | 0
  Dyspepsia: Subject did not experience this treatment-related toxicity | 10
  Gastroesophageal Reflux disease: Grade 1 (CTCAE v4) | 1
  Gastroesophageal Reflux disease: Grade 2 (CTCAE v4) | 0
  Gastroesophageal Reflux disease: Grade 3 (CTCAE v4) | 0
  Gastroesophageal Reflux disease: Subject did not experience this treatment-related toxicity | 10
  Gastrointestinal disorders - other, specify: Grade 1 (CTCAE v4) | 1
  Gastrointestinal disorders - other, specify: Grade 2 (CTCAE v4) | 1
  Gastrointestinal disorders - other, specify: Grade 3 (CTCAE v4) | 0
  Gastrointestinal disorders - other, specify: Subject did not experience this treatment-related toxicity | 9
  Mucositis oral: Grade 1 (CTCAE v4) | 1
  Mucositis oral: Grade 2 (CTCAE v4) | 2
  Mucositis oral: Grade 3 (CTCAE v4) | 0
  Mucositis oral: Subject did not experience this treatment-related toxicity | 8
  Nausea: Grade 1 (CTCAE v4) | 2
  Nausea: Grade 2 (CTCAE v4) | 0
  Nausea: Grade 3 (CTCAE v4) | 0
  Nausea: Subject did not experience this treatment-related toxicity | 9
  Oral pain: Grade 1 (CTCAE v4) | 0
  Oral pain: Grade 2 (CTCAE v4) | 1
  Oral pain: Grade 3 (CTCAE v4) | 0
  Oral pain: Subject did not experience this treatment-related toxicity | 10
  Fatigue: Grade 1 (CTCAE v4) | 3
  Fatigue: Grade 2 (CTCAE v4) | 0
  Fatigue: Grade 3 (CTCAE v4) | 0
  Fatigue: Subject did not experience this treatment-related toxicity | 8
  Fever: Grade 1 (CTCAE v4) | 0
  Fever: Grade 2 (CTCAE v4) | 0
  Fever: Grade 3 (CTCAE v4) | 1
  Fever: Subject did not experience this treatment-related toxicity | 10
  Paronychia: Grade 1 (CTCAE v4) | 2
  Paronychia: Grade 2 (CTCAE v4) | 2
  Paronychia: Grade 3 (CTCAE v4) | 0
  Paronychia: Subject did not experience this treatment-related toxicity | 7
  Alanine aminotransferase increased: Grade 1 (CTCAE v4) | 3
  Alanine aminotransferase increased: Grade 2 (CTCAE v4) | 2
  Alanine aminotransferase increased: Grade 3 (CTCAE v4) | 0
  Alanine aminotransferase increased: Subject did not experience this treatment-related toxicity | 6
  Aspartate aminotransferase increased: Grade 1 (CTCAE v4) | 4
  Aspartate aminotransferase increased: Grade 2 (CTCAE v4) | 0
  Aspartate aminotransferase increased: Grade 3 (CTCAE v4) | 0
  Aspartate aminotransferase increased: Subject did not experience this treatment-related toxicity | 7
  Electrocardiogram QT corrected interval prolonged: Grade 1 (CTCAE v4) | 1
  Electrocardiogram QT corrected interval prolonged: Grade 2 (CTCAE v4) | 0
  Electrocardiogram QT corrected interval prolonged: Grade 3 (CTCAE v4) | 0
  Electrocardiogram QT corrected interval prolonged: Subject did not experience this treatment-related toxicity | 10
  Neutrophil count decreased: Grade 1 (CTCAE v4) | 2
  Neutrophil count decreased: Grade 2 (CTCAE v4) | 0
  Neutrophil count decreased: Grade 3 (CTCAE v4) | 0
  Neutrophil count decreased: Subject did not experience this treatment-related toxicity | 9
  Weight gain: Grade 1 (CTCAE v4) | 1
  Weight gain: Grade 2 (CTCAE v4) | 0
  Weight gain: Grade 3 (CTCAE v4) | 0
  Weight gain: Subject did not experience this treatment-related toxicity | 10
  Anorexia: Grade 1 (CTCAE v4) | 1
  Anorexia: Grade 2 (CTCAE v4) | 0
  Anorexia: Grade 3 (CTCAE v4) | 0
  Anorexia: Subject did not experience this treatment-related toxicity | 10
  Hypomagnesemia: Grade 1 (CTCAE v4) | 1
  Hypomagnesemia: Grade 2 (CTCAE v4) | 0
  Hypomagnesemia: Grade 3 (CTCAE v4) | 0
  Hypomagnesemia: Subject did not experience this treatment-related toxicity | 10
  Hyponatremia: Grade 1 (CTCAE v4) | 1
  Hyponatremia: Grade 2 (CTCAE v4) | 0
  Hyponatremia: Grade 3 (CTCAE v4) | 0
  Hyponatremia: Subject did not experience this treatment-related toxicity | 10
  Metabolism and nutrition disorders - other, specify: Grade 1 (CTCAE v4) | 1
  Metabolism and nutrition disorders - other, specify: Grade 2 (CTCAE v4) | 0
  Metabolism and nutrition disorders - other, specify: Grade 3 (CTCAE v4) | 0
  Metabolism and nutrition disorders - other, specify: Subject did not experience this treatment-related toxicity | 10
  Arthralgia: Grade 1 (CTCAE v4) | 1
  Arthralgia: Grade 2 (CTCAE v4) | 0
  Arthralgia: Grade 3 (CTCAE v4) | 0
  Arthralgia: Subject did not experience this treatment-related toxicity | 10
  Myalgia: Grade 1 (CTCAE v4) | 3
  Myalgia: Grade 2 (CTCAE v4) | 0
  Myalgia: Grade 3 (CTCAE v4) | 0
  Myalgia: Subject did not experience this treatment-related toxicity | 8
  Renal and urinary disorders - other, specify: Grade 1 (CTCAE v4) | 1
  Renal and urinary disorders - other, specify: Grade 2 (CTCAE v4) | 0
  Renal and urinary disorders - other, specify: Grade 3 (CTCAE v4) | 0
  Renal and urinary disorders - other, specify: Subject did not experience this treatment-related toxicity | 10
  Erectile dysfunction: Grade 1 (CTCAE v4) | 1
  Erectile dysfunction: Grade 2 (CTCAE v4) | 0
  Erectile dysfunction: Grade 3 (CTCAE v4) | 0
  Erectile dysfunction: Subject did not experience this treatment-related toxicity | 10
  Vaginal pain: Grade 1 (CTCAE v4) | 1
  Vaginal pain: Grade 2 (CTCAE v4) | 0
  Vaginal pain: Grade 3 (CTCAE v4) | 0
  Vaginal pain: Subject did not experience this treatment-related toxicity | 10
  Cough: Grade 1 (CTCAE v4) | 0
  Cough: Grade 2 (CTCAE v4) | 1
  Cough: Grade 3 (CTCAE v4) | 0
  Cough: Subject did not experience this treatment-related toxicity | 10
  Dyspnea: Grade 1 (CTCAE v4) | 0
  Dyspnea: Grade 2 (CTCAE v4) | 1
  Dyspnea: Grade 3 (CTCAE v4) | 0
  Dyspnea: Subject did not experience this treatment-related toxicity | 10
  Epistaxis: Grade 1 (CTCAE v4) | 1
  Epistaxis: Grade 2 (CTCAE v4) | 0
  Epistaxis: Grade 3 (CTCAE v4) | 0
  Epistaxis: Subject did not experience this treatment-related toxicity | 10
  Pneumonitis: Grade 1 (CTCAE v4) | 0
  Pneumonitis: Grade 2 (CTCAE v4) | 1
  Pneumonitis: Grade 3 (CTCAE v4) | 0
  Pneumonitis: Subject did not experience this treatment-related toxicity | 10
  Sore throat: Grade 1 (CTCAE v4) | 0
  Sore throat: Grade 2 (CTCAE v4) | 1
  Sore throat: Grade 3 (CTCAE v4) | 0
  Sore throat: Subject did not experience this treatment-related toxicity | 10
  Alopecia: Grade 1 (CTCAE v4) | 1
  Alopecia: Grade 2 (CTCAE v4) | 1
  Alopecia: Grade 3 (CTCAE v4) | 0
  Alopecia: Subject did not experience this treatment-related toxicity | 9
  Bullous dermatitis: Grade 1 (CTCAE v4) | 0
  Bullous dermatitis: Grade 2 (CTCAE v4) | 1
  Bullous dermatitis: Grade 3 (CTCAE v4) | 0
  Bullous dermatitis: Subject did not experience this treatment-related toxicity | 10
  Dry skin: Grade 1 (CTCAE v4) | 4
  Dry skin: Grade 2 (CTCAE v4) | 1
  Dry skin: Grade 3 (CTCAE v4) | 0
  Dry skin: Subject did not experience this treatment-related toxicity | 6
  Erythema multiforme: Grade 1 (CTCAE v4) | 2
  Erythema multiforme: Grade 2 (CTCAE v4) | 0
  Erythema multiforme: Grade 3 (CTCAE v4) | 0
  Erythema multiforme: Subject did not experience this treatment-related toxicity | 9
  Pain of skin: Grade 1 (CTCAE v4) | 1
  Pain of skin: Grade 2 (CTCAE v4) | 1
  Pain of skin: Grade 3 (CTCAE v4) | 0
  Pain of skin: Subject did not experience this treatment-related toxicity | 9
  Pruritis: Grade 1 (CTCAE v4) | 4
  Pruritis: Grade 2 (CTCAE v4) | 1
  Pruritis: Grade 3 (CTCAE v4) | 0
  Pruritis: Subject did not experience this treatment-related toxicity | 6
  Rash acneiform: Grade 1 (CTCAE v4) | 5
  Rash acneiform: Grade 2 (CTCAE v4) | 2
  Rash acneiform: Grade 3 (CTCAE v4) | 0
  Rash acneiform: Subject did not experience this treatment-related toxicity | 4
  Rash maculo-papular: Grade 1 (CTCAE v4) | 3
  Rash maculo-papular: Grade 2 (CTCAE v4) | 2
  Rash maculo-papular: Grade 3 (CTCAE v4) | 3
  Rash maculo-papular: Subject did not experience this treatment-related toxicity | 3
  Scalp pain: Grade 1 (CTCAE v4) | 1
  Scalp pain: Grade 2 (CTCAE v4) | 0
  Scalp pain: Grade 3 (CTCAE v4) | 0
  Scalp pain: Subject did not experience this treatment-related toxicity | 10
  Skin/subcutaneous tissue disorders - other, specify: Grade 1 (CTCAE v4) | 3
  Skin/subcutaneous tissue disorders - other, specify: Grade 2 (CTCAE v4) | 1
  Skin/subcutaneous tissue disorders - other, specify: Grade 3 (CTCAE v4) | 0
  Skin/subcutaneous tissue disorders - other, specify: Subject did not experience this treatment-related toxicity | 7

ADVERSE EVENTS:
Time Frame: Adverse events are collected from informed consent until 30 days after the end of treatment (maximum 4 years and 5 months). Patients were monitored for survival up to 6 years.
Arm/Group | EGF816 + Gefitinib
All-Cause Mortality (participants affected / at risk) | 4/11
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGF816 + Gefitinib (N=11)
Fever (General disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGF816 + Gefitinib (N=11)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 5
Allergic reaction (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bloating (Gastrointestinal disorders) | 1
Blood and lymphatic system disorders - Other, specify: Hyperlipidemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify: Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Cardiac disorders - Other, specify: heartburn (Cardiac disorders) | 1
Cardiac disorders - Other, specify: Papillary Fibroelastoma of the Heart (Cardiac disorders) | 1
Cardiac disorders - Other, specify: Prolonged QT (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 3
Cholesterol high (Investigations) | 2
Cognitive disturbance (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Creatinine increased (Investigations) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 2
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Electrocardiogram QT corrected interval prolonged (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Eye pain (Eye disorders) | 1
Fatigue (General disorders) | 6
Fever (General disorders) | 5
Floaters (Eye disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify: mouth sores (Gastrointestinal disorders) | 2
General disorders and administration site conditions - Other, specify: Lisinopril allergy (General disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Immune system disorders - Other, specify: Environmental Allergy (Immune system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Metabolism and nutrition disorders - Other, specify: Decrease Appetite (Metabolism and nutrition disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify: Right Knee Strain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Right hip discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: numbness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify: Sciatica (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Neck edema (General disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neutrophil count decreased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 3
Paresthesia (Nervous system disorders) | 1
Paronychia (Infections and infestations) | 4
Pericardial tamponade (Cardiac disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Renal and urinary disorders - Other, specify: Dysuria (Renal and urinary disorders) | 1
Respiratory, thoracic and mediastinal disorders - other, specify: Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders: other: Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Blister on right toe (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Angular Cheilitis (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Tenderness and redness of left fourth finger (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: cracks of the fingertips (Skin and subcutaneous tissue disorders) | 1
Skin/subcutaneous tissue disorders; Other, specify: Hypersensitivity (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Syncope (Nervous system disorders) | 1
Vaginal Pain (Reproductive system and breast disorders) | 1
Weight gain (Investigations) | 1

LIMITATIONS AND CAVEATS:
While the original sample size was planned to be 36 patients, only 11 patients were enrolled, as the study was terminated early due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT03292133/Prot_SAP_000.pdf